CLINICAL TRIAL: NCT02609178
Title: Comparative Evaluation of Different Occlusal Surface Designs of Artificial Crown
Brief Title: Basic Study of Fabricating Biomorphic Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Ji-hua Chen, Dean, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-REV-2015039
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-06

CONDITIONS: Dental Crown; Prosthesis
Keywords: artificial crown; biomorphic; functional generated path; muscle-action theory; anatomic theory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FGP design (FGP, AVR) (Experimental): use functional generated path to execute different occlusal surface designs of the artificial crown and evaluate its efficacy
  Interventions: Procedure: FGP; Procedure: AVR
- conventional design (CON) (No Intervention): use conventional method to execute different occlusal surface designs of the artificial crown and evaluate its efficacy

INTERVENTIONS:
Procedure: FGP — To execute FGP technique, the occlusal surface of the interim should be back cut to leave at least 1mm occlusal space. Then apply the recording resin. Ask the subjects to close the mouth to maximum intercuspal position then perform right lateral, left lateral and protrusive movements in succession ending in maximum intercuspation position. Excessive resin then should be trimmed off and Bausch articulating paper would be used to mark the intercuspal contacts. Zinc oxide is then applied to check eccentric occlusion, trimmed off resin if there're interferences. Then the interim would be used as a copy to design the occlusal surface of the crown. (CAD/CAM)
  Other Names: general
  Arms: FGP design (FGP, AVR)
Procedure: AVR — the crowns in this group would be designed by setting virtual articulator to average mode (CAD/CAM)
  Other Names: average value
  Arms: FGP design (FGP, AVR)

SUMMARY:
The purpose of this study is to compare among different designs of the occlusal surface of artificial crowns, trying to determine a guidance of fabricating artificial crowns with better mimesis of the original tooth crown in terms of morphology.

DETAILED DESCRIPTION:
For occlusal surface design, each subject would be given 3 crowns using different fabricating guidance -- the FGP technique(FGP),the average setting technique(AVR) and conventional technique(CON), separately. Upon baseline visit, general tooth preparation procedures would be performed, including impression taking before and after treatment and tooth preparation. Sometimes photo taking is needed. On try-in visit, subjects would be ask to fill in questionaires(Likert's scale) and the adjusting time for each crown would be recorded. Moreover, t-scan would be used to assess the occlusal equilibrium. All in all, including adjusting visit for FGP, the subjects have to visit the clinic for 3 times which would take them 3-week time.

The Institutional Board(IRB) of the Stomatological Hospital of Fourth Military Medical University(FMMU) would be in supervision of the whole study and is responsible for the quality assurance plan, data check and source data verification.

Subject recruitment would done within those patients visit the department of prosthodontics of the Stomatological Hospital of FMMU and have an interest towards this study. One clinician would be appointed to enroll the subjects according to the standards. To avoid errors, all the examinations done in the study shall be accomplished by the same clinician and the crowns fabricated in the study shall be designed by the same technician. The clinician and the technician participated would receive adequate training before the study to ensure their performance. Every subject in the study should assign informed consents at the beginning of the study and establish case report forms(CRFs). During the study, if adverse events(such as crown chipping, crown dropping or iatrogenic gingivitis, etc) happen, subjects are required to contact the investigator within 24 hours; and the investigator should then report to the IRB within 24 hours. Following treatment or compensation would be done according to the clauses stated in the informed consent signed by the subjects.

The whole study needs subjects in total. During the study, subjects have their own right to quit the study at any time if they have discussed with the investigator in advance. These subjects then are deemed as "unavailable". If subjects don't contact the investigator and quit the study(the investigators can't contact them within the follow-up period), their records then are deemed as "missing".

All the information collected in the study would be protected and only be used within this study. The statistical analysis of this study would be processed with the aid of the department of statistics of FMMU.

ELIGIBILITY:
Inclusion Criteria:

* single crown restoration needed in posterior quadrants
* the antagonist of the abutment tooth is purely natural or received minimum restorations that does not change its morphology too much
* no orthodontic treatment history
* stable occlusion
* no parafunctional movements existed

Exclusion Criteria:

* sequential crown restorations needed
* the morphology of the antagonist of the abutment tooth has been largely changed by previous treatment
* no contact exists between the abutment tooth and its antagonist
* orthodontic treatment history
* unstable occlusion
* existed parafunctional movements
* participated in other clinical studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jihua Chen, PhD, Study Chair — Stomatological Hospital of FMMU
Locations (1):
- Stomatological Hospital of Fourth Military Medical University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mehl A. A new concept for the integration of dynamic occlusion in the digital construction process. Int J Comput Dent. 2012;15(2):109-23. English, German. PMID 22891415
- [Background] Ikeda A, Miura H, Okada D, Tokuda A, Shinogaya T. The effect of occlusal contacts on adjacent tooth. J Med Dent Sci. 2005 Dec;52(4):195-202. PMID 16669453
- [Background] Alhouri N, Watts DC, McCord JF, Smith PW. Mathematical analysis of tooth and restoration contour using image analysis. Dent Mater. 2004 Nov;20(9):893-9. doi: 10.1016/j.dental.2004.06.003. PMID 15451245
- [Background] Vasconcelos FS, Neves AC, Silva-Concilio LR, Cunha LG, Rode Sde M. Influence of anatomic reference on the buccal contour of prosthetic crowns. Braz Oral Res. 2009 Jul-Sep;23(3):230-5. doi: 10.1590/s1806-83242009000300002. PMID 19893955
- [Background] Kohal RJ, Gerds T, Strub JR. Effect of different crown contours on periodontal health in dogs. Clinical results. J Dent. 2003 Aug;31(6):407-13. doi: 10.1016/s0300-5712(03)00070-8. PMID 12878023
- [Background] Takada J, Ono T, Miyamoto JJ, Yokota T, Moriyama K. Association between intraoral pressure and molar position and inclination in subjects with facial asymmetry. Eur J Orthod. 2011 Jun;33(3):243-9. doi: 10.1093/ejo/cjq060. Epub 2010 Sep 9. PMID 20829312
- [Background] Olthoff L, Meijer I, de Ruiter W, Bosman F, van der Zel J. Effect of virtual articulator settings on occlusal morphology of CAD/CAM restorations. Int J Comput Dent. 2007 Apr;10(2):171-85. English, German. PMID 17899892
- [Background] Memon S. A Comparative Evaluation of the Effect of Double Casting Technique Using Functionally Generated Path and Conventional Single Casting with Respect to Functional Articulation, Patient Satisfaction and Chair Side Time, in Single Unit Molar Teeth: An In Vivo Study. J Indian Prosthodont Soc. 2014 Dec;14(Suppl 1):119-25. doi: 10.1007/s13191-014-0379-6. Epub 2014 Jul 10. PMID 26199501
- [Background] Curtis SR. Functionally generated paths for ceramometal restorations. J Prosthet Dent. 1999 Jan;81(1):33-6. doi: 10.1016/s0022-3913(99)70232-5. PMID 9878972
- [Background] Wiklund L, Rossi F, Strata P, van der Want JJ. The rat olivocerebellar system visualized in detail with anterograde PHA-L tracing technique, and sprouting of climbing fibers demonstrated after subtotal olivary lesions. Eur J Morphol. 1990;28(2-4):256-67. PMID 2245134
- [Background] Ender A, Mormann WH, Mehl A. Efficiency of a mathematical model in generating CAD/CAM-partial crowns with natural tooth morphology. Clin Oral Investig. 2011 Apr;15(2):283-9. doi: 10.1007/s00784-010-0384-z. Epub 2010 Feb 9. PMID 20143242
- [Background] Becker CM, Kaldahl WB. Current theories of crown contour, margin placement, and pontic design. 1981. J Prosthet Dent. 2005 Feb;93(2):107-15. doi: 10.1016/j.prosdent.2004.11.005. No abstract available. PMID 15674218
- [Background] Hazen SP, Osborne JW. Relationship of operative dentistry to periodontal health. Dent Clin North Am. 1967 Mar:245-54. No abstract available. PMID 5225601
- [Background] Yuodelis RA, Weaver JD, Sapkos S. Facial and lingual contours of artificial complete crown restorations and their effects on the periodontium. J Prosthet Dent. 1973 Jan;29(1):61-6. doi: 10.1016/0022-3913(73)90140-6. No abstract available. PMID 4564800
- [Background] Koidis PT, Burch JG, Melfi RC. Clinical crown contours: contemporary view. J Am Dent Assoc. 1987 Jun;114(6):792-5. doi: 10.14219/jada.archive.1987.0189. PMID 3301975
- [Background] Parkinson CF. Excessive crown contours facilitate endemic plaque niches. J Prosthet Dent. 1976 Apr;35(4):424-9. doi: 10.1016/0022-3913(76)90010-x. PMID 1062611
- [Background] Cho SH, Chang WG. Mirror-image anterior crown fabrication with computer-aided design and rapid prototyping technology: a clinical report. J Prosthet Dent. 2013 Feb;109(2):75-8. doi: 10.1016/S0022-3913(13)60018-9. PMID 23395331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the participants were enrolled from the Department of Prosthodontics, Stomatological Hospital of Fourth Military Medical University between December 2015 and March 2016.
Pre-assignment Details: 17 patients assessed for eligibility, 5 of them were excluded for not meeting inclusion criteria. 12 participants recruited; 10 screened.
Groups:
- FGP First, Then AVR, Then CON: Tried in the artificial crowns for the same participant as the following sequence: FGP, AVR, CON, a 5-min washout period would be given between each crown.
- FGP First, Then CON, Then AVR: Tried in the artificial crowns for the same participant as the following sequence: FGP, CON, AVR, a 5-min washout period would be given between each crown.
- AVR First, Then FGP, Then CON: Tried in the artificial crowns for the same participant as the following sequence: AVR, FGP, CON, a 5-min washout period would be given between each crown.
- AVR First, Then CON, Then FGP: Tried in the artificial crowns for the same participant as the following sequence: AVR, CON, FGP, a 5-min washout period would be given between each crown.
- CON First, Then FGP, Then AVR: Tried in the artificial crowns for the same participant as the following sequence: CON, FGP, AVR, a 5-min washout period would be given between each crown.
- CON First, Then AVR, Then FGP: Tried in the artificial crowns for the same participant as the following sequence: CON, AVR, FGP, a 5-min washout period would be given between each crown.
Period: First Crown
Arm/Group | FGP First, Then AVR, Then CON | FGP First, Then CON, Then AVR | AVR First, Then FGP, Then CON | AVR First, Then CON, Then FGP | CON First, Then FGP, Then AVR | CON First, Then AVR, Then FGP
Started | 0 | 1 | 6 | 3 | 0 | 2
Completed | 0 | 1 | 5 | 2 | 0 | 2
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0 | 0
Period: 5-minute Washout Time
Arm/Group | FGP First, Then AVR, Then CON | FGP First, Then CON, Then AVR | AVR First, Then FGP, Then CON | AVR First, Then CON, Then FGP | CON First, Then FGP, Then AVR | CON First, Then AVR, Then FGP
Started | 0 | 1 | 5 | 2 | 0 | 2
Completed | 0 | 1 | 5 | 2 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Crown
Arm/Group | FGP First, Then AVR, Then CON | FGP First, Then CON, Then AVR | AVR First, Then FGP, Then CON | AVR First, Then CON, Then FGP | CON First, Then FGP, Then AVR | CON First, Then AVR, Then FGP
Started | 0 | 1 | 5 | 2 | 0 | 2
Completed | 0 | 1 | 5 | 2 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: 5-minute Washout Time
Arm/Group | FGP First, Then AVR, Then CON | FGP First, Then CON, Then AVR | AVR First, Then FGP, Then CON | AVR First, Then CON, Then FGP | CON First, Then FGP, Then AVR | CON First, Then AVR, Then FGP
Started | 0 | 1 | 5 | 2 | 0 | 2
Completed | 0 | 1 | 5 | 2 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Crown
Arm/Group | FGP First, Then AVR, Then CON | FGP First, Then CON, Then AVR | AVR First, Then FGP, Then CON | AVR First, Then CON, Then FGP | CON First, Then FGP, Then AVR | CON First, Then AVR, Then FGP
Started | 0 | 1 | 5 | 2 | 0 | 2
Completed | 0 | 1 | 5 | 2 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Occlusal Surface Design: use computer-aided design and computer-aided manufacturing technique (CAD/CAM) to execute different occlusal surface designs of the artificial crown, including FGP design (FGP and AVR) and conventional design (CON), and evaluate their efficacy, separately
Arm/Group | Occlusal Surface Design
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  China | 12

OUTCOME MEASURES:

1. Primary Outcome: △OT Value
Description: Occlusion time (OT) is defined as the time from the first contact of occluding teeth to maximum intercuspation. OT is directly related with patients' occlusal contact pattern; and some have considered it as a capable description of occlusion.
  In the study, the OT value of each crown would be assessed before try-in (baseline) and immediately after try-in using T-scan (FGP, AVR, CON). Try-in procedure would be finished by the same clinician.
  △OT was calculated for minimizing individual difference among participants. The equation for △OT was:△OT(FGP/ AVR/ CON)= OT (FGP/ AVR/ CON)-OT(baseline)
Time Frame: 2 weeks(plus or minus 7 days) after tooth preparation
Population: Including participants who tried in all of the three differently designed artificial crowns.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- FGP Designed Surface: The occlusal surface of the artificial crown was designed by FGP technique.
- AVR Designed Surface: The occlusal surface of the artificial crown was designed by setting the virtual articulator at average values, that is, 30° for the angles of the sagittal condyle and 15° for the lateral Bennett angle, and 30° for the incisal path, respectively.
- CON Designed Surface: The occlusal surface of the artificial crown was fabricated based on the technicians' experience.
Arm/Group | FGP Designed Surface | AVR Designed Surface | CON Designed Surface
Number analyzed (Participants) | 10 | 10 | 10
seconds | 0.07 (0.09) | 0.13 (0.06) | 0.22 (0.10)
Statistical Analysis 1: Comparison: FGP Designed Surface vs AVR Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Using G*power 3.1.7, setting α at 0.05, (1- β) at 0.8, the number of the subjects enrolled could reach the actual power as 0.8; p = 0.003, ANOVA — Alpha value was set at 0.05
Statistical Analysis 2: Comparison: FGP Designed Surface vs AVR Designed Surface; Test type: Non-Inferiority or Equivalence — stated above in statistical analysis 1; p = 0.366, Tukey's multiple comparison test — Alpha value was set at 0.05
Statistical Analysis 3: Comparison: FGP Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.002, Tukey's multiple comparison test — Alpha value was set at 0.05
Statistical Analysis 4: Comparison: AVR Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.054, Tukey's multiple comparison test — Alpha value was set at 0.05

2. Secondary Outcome: Occlusal Adjusting Time for Crowns
Description: Try-in procedure would be finished by the same clinician. The occlusal adjusting time would be counted using a timer and recorded.
Time Frame: 2 weeks(plus or minus 7 days) after tooth preparation
Population: Including participants who tried in all of the three differently designed artificial crowns.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | FGP Designed Surface | AVR Designed Surface | CON Designed Surface
Number analyzed (Participants) | 10 | 10 | 10
minutes | 5.4 (3.8) | 6.1 (4.8) | 12.6 (5.3)
Statistical Analysis 1: Comparison: FGP Designed Surface vs AVR Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.006, Kruskal-Wallis — alpha value was set at 0.05
Statistical Analysis 2: Comparison: FGP Designed Surface vs AVR Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistic analysis 1; p = 0.739, Wilcoxon (Mann-Whitney) — Alpha value was set at 0.05
Statistical Analysis 3: Comparison: FGP Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.03, Wilcoxon (Mann-Whitney) — Alpha value was set at 0.05
Statistical Analysis 4: Comparison: AVR Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.009, Wilcoxon (Mann-Whitney) — Alpha value was set at 0.05

3. Secondary Outcome: Likert's Scale
Description: The questionaire was designed to evaluate participants' feeling towards the occlusal interference. It would be given to the subject after immediately try-in the crowns. In the questionaire:
  Score 0 = No interference (feel comfortable while biting on the artificial crown) Score 1 = Moderate interference(could feel the artificial crown is higher when biting on the artificial crown, but when firmly clenched, the upper teeth could bite on the lower ones) Score 2 = High interference(the artificial teeth is higher that the upper teeth couldn't bite on all the lower teeth when firmly clenched)
Time Frame: 2 weeks(plus or minus 7 days) after tooth preparation
Population: Including participants who tried in all of the three differently designed artificial crowns.
Measure: Number; unit: participants
Arm/Group | FGP Designed Surface | AVR Designed Surface | CON Designed Surface
Number analyzed (Participants) | 10 | 10 | 10
participants
  Score 0 | 4 | 3 | 0
  Score 1 | 5 | 5 | 1
  Score 2 | 1 | 2 | 9
Statistical Analysis 1: Comparison: FGP Designed Surface; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.001, Kruskal-Wallis — alpha value was set at 0.05
Statistical Analysis 2: Comparison: FGP Designed Surface vs AVR Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.579, Wilcoxon (Mann-Whitney) — Alpha value was set at 0.05
Statistical Analysis 3: Comparison: FGP Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.001, Wilcoxon (Mann-Whitney) — Alpha value was set at 0.05
Statistical Analysis 4: Comparison: AVR Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.002, Wilcoxon (Mann-Whitney) — Alpha value was set at 0.05

4. Primary Outcome: △DT Value
Description: Disocclusion time (DT) is defined as the time from maximum intercuspation to complete disocclusion during lateral movement. DT related tooth contacts with muscle activity. Abnormities in DT would result in change of muscle activity, thus facilitate the occurrence of temporomandibular joint disorders.
  In the study, the DT value of each crown would be assessed before try-in (baseline) and immediately after try-in using T-scan (FGP, AVR, CON). Try-in procedure would be finished by the same clinician.
  △DT was calculated for minimizing individual difference among participants. The equation for △DT was: △DT(FGP/ AVR/ CON)= DT (FGP/ AVR/ CON)-DT(baseline)
Time Frame: 2 weeks(plus or minus 7 days) after tooth preparation
Population: Including participants who tried in all of the three differently designed artificial crowns.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | FGP Designed Surface | AVR Designed Surface | CON Designed Surface
Number analyzed (Participants) | 10 | 10 | 10
seconds | 0.09 (0.51) | 0.49 (0.58) | 1.02 (0.69)
Statistical Analysis 1: Comparison: FGP Designed Surface vs AVR Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.007, ANOVA — alpha value was set at 0.05
Statistical Analysis 2: Comparison: FGP Designed Surface vs AVR Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.308, Tukey's multiple comparison test — Alpha value was set at 0.05
Statistical Analysis 3: Comparison: FGP Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.005, Tukey's multiple comparison test — Alpha value was set at 0.05
Statistical Analysis 4: Comparison: AVR Designed Surface vs CON Designed Surface; Test type: Non-Inferiority or Equivalence — Stated above in statistical analysis 1; p = 0.141, Tukey's multiple comparison test — Alpha value was set at 0.05

ADVERSE EVENTS:
Time Frame: 3 months
Description: Serious Adverse Events were not collected.
Arm/Group | Occlusal Surface Design
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes